CLINICAL TRIAL: NCT02187120
Title: A Multi-centre Randomised, Double-blinded, Placebo-controlled Trial of Pre-hospital Treatment With Tranexamic Acid for Severely Injured Patients at Risk of Acute Traumatic Coagulopathy.
Brief Title: Pre-hospital Anti-fibrinolytics for Traumatic Coagulopathy and Haemorrhage (The PATCH Study)
Acronym: PATCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Russell Gruen, Professor of Surgery and Public Health, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APP1044894; U1111-1160-6738 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Wounds and Injuries; Acute Coagulopathy
Keywords: Wounds and Injuries; Acute Coagulopathy; Tranexamic Acid; Emergency Medical Services
MeSH Terms: conditions — Wounds and Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): As soon as possible after injury, emergency medical services clinicians will administer 1g Tranexamic Acid (10ml ampoule containing 100mg/ml Tranexamic Acid in water for injection) delivered intravenously using a slow push of the syringe.
  As soon as possible after the patient arrives at hospital, clinicians will administer 1g Tranexamic acid (10ml ampoule containing 100mg/ml Tranexamic Acid in water for injection) added to up to one litre 0.9%w/v Sodium Chloride and the entire volume infused intravenously over 8 hours.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): As soon as possible after injury, emergency medical services clinicians will administer a 10ml ampoule containing 0.9%w/v Sodium Chloride via intravenous injection using a slow push of the syringe (ampoules containing Sodium Chloride appear identical to the ampoules containing Tranexamic Acid).
  As soon as possible after the patient arrives at hospital, clinicians will administer a second 10 ml ampoule containing 0.9%w/v Sodium Chloride added to up to one litre 0.9%w/v Sodium Chloride and the entire volume infused intravenously over 8 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid is a synthetic lysine derivative that inhibits fibrinolysis by blocking the lysine binding sites on plasminogen therefore inhibiting the conversion of plasminogen to plasmin. Intravenous injection of 1g Tranexamic Acid will be administered in the pre-hospital setting followed by 1g Tranexamic Acid infused intravenously over 8 hours initiated in the hospital emergency department.
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to determine whether giving severely injured adults a drug called tranexamic acid (TXA) as soon as possible after injury will improve their chances of survival and their level of recovery at six months.

After severe injury, a person may have uncontrolled bleeding that places them at high risk of bleeding to death. Coagulation (the formation of blood clots) is an important process in the body that helps to control blood loss. Up to a quarter of people that are severely injured have a condition called acute traumatic coagulopathy. This condition affects coagulation and results in the break down of blood clots (fibrinolysis) that can lead to increased blood loss and an increased risk of dying.

TXA is an anti-fibrinolytic drug that might help to reduce the effects of acute traumatic coagulopathy by preventing blood clots from breaking down and helping to control bleeding. In Australia, TXA is approved for use by the Therapeutic Goods Administration (TGA) to reduce blood loss or the need for blood transfusion in patients undergoing surgery (i.e. cardiac surgery, knee or hip arthroplasty). Recent evidence from a large clinical trial (CRASH-2) showed early treatment with TXA reduced the risk of death in severely injured patients, however the majority of patients involved in the study were injured in countries where prehospital care is limited and rapid access to lifesaving treatments is limited compared to that available in countries like Australia and New Zealand. It is unclear whether TXA will reduce the risk of death to the same degree when it is given alongside other lifesaving treatments that are available to patients soon after injury in these countries.

The hypothesis is that TXA given early to injured patients who are at risk of acute traumatic coagulopathy and who are treated in countries with systems providing advanced trauma care reduces mortality and improves recovery at 6-months after injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (estimated age 18 years or older)
* Injured through any mechanism
* Coagulopathy of severe trauma (COAST) score of 3 points or greater
* First dose of study drug can be administered within three hours of injury
* Patients to be transported to a participating trauma centre

COAST score

* Entrapment (ie in vehicle) [Yes = 1, No = 0]
* Systolic blood pressure [<90 mmHg = 2, <100 mmHg = 1, ≥100 mmHg = 0]
* Temperature [<32℃ =2, <35℃ = 1, ≥35℃ = 0]
* Major chest injury likely to require intervention (e.g. decompression, chest tube) [Yes = 1, No = 0]
* Likely intra-abdominal or pelvic injury [Yes = 1, No = 0]

Exclusion Criteria:

* Suspected pregnancy
* Nursing home residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a favourable outcome (moderate disability or good recovery, GOSE scores 5-8) compared to those who have died (GOSE 1), or have severe disability (GOSE 2-4). | 6 months

SECONDARY OUTCOMES:
Units of blood products used (red blood cells, plasma, platelets, prothrombin complex concentrate, fibrinogen, Factor VIIa, cryoprecipitate) | 24 hours
Coagulation assessed using the international normalised ratio (INR) | Immediately upon patient arrival to hospital
Coagulation assessed using the international normalised ratio (INR) | At the end of 8 hour infusion of study drug
Coagulation assessed using the international normalised ratio (INR) | 24 hours after pre-hospital dose of study drug
Coagulation assessed by activated partial thromboplastin time (APTT) | Immediately upon patient arrival to hospital
Coagulation assessed by activated partial thromboplastin time (APTT) | At the end of 8 hour infusion of study drug
Coagulation assessed by activated partial thromboplastin time (APTT) | 24 hours after pre-hospital dose of study drug
Platelet count | Immediately upon patient arrival to hospital
Platelet count | At the end of 8 hour infusion of study drug
Platelet count | 24 hours after pre-hospital dose of study drug
Vascular occlusive events (myocardial infarction, stroke, deep venous thrombosis (DVT), pulmonary embolus (PE)) | Hospital discharge (or up to 28 days in hospital)
Ventilator-free days | 28 days
Mortality | 24 hours
Mortality | 28 days
Mortality | 6 months
Proportion of deaths due to bleeding, vascular occlusion (pulmonary embolus, stroke, acute myocardial infarction), multi-organ failure, or head injury | 24 hours
Proportion of deaths due to bleeding, vascular occlusion (pulmonary embolus, stroke, acute myocardial infarction), multi-organ failure, or head injury | 28 days
Proportion of deaths due to bleeding, vascular occlusion (pulmonary embolus, stroke, acute myocardial infarction), multi-organ failure, or head injury | 6 months
Cumulative incidence of sepsis | Hospital discharge (or up to 28 days in hospital)
Quality of life measured using WHODAS 2.0 | 6 months
Quality of life measured using the EuroQOL 5 dimensions questionnaire (EQ-5D) | 6 months
Number of participants with serious adverse events | hospital discharge (or up to 28 days in hospital)
Coagulation assessed by fibrinogen | Immediately upon patient arrival to hospital
Coagulation assessed by fibrinogen | At the end of 8 hour infusion of study drug
Coagulation assessed by fibrinogen | 24 hours after pre-hospital dose of study drug

OTHER OUTCOMES:
Blood lactate concentration | Immediately upon patient arrival to hospital
Laboratory analysis of fibrinolytic activity | At the end of 8 hour infusion of study drug
Laboratory analysis of fibrinolytic activity | 24 hours after first (prehospital) dose of study drug
Laboratory analysis of plasmin/anti-plasmin complexes | At the end of 8 hour infusion of study drug
Laboratory analysis of plasmin/anti-plasmin complexes | 24 hours after first (pre-hospital) dose of study drug
Laboratory analysis of tissue type plasminogen activator (tPA) | At the end of 8 hour infusion of study drug
Laboratory analysis of tissue type plasminogen activator (tPA) | 24 hours after first (pre-hospital) dose of study drug
Laboratory analysis of plasminogen activator inhibitor 1 (PAI-1) | At the end of 8 hour infusion of study drug
Laboratory analysis of plasminogen activator inhibitor 1 (PAI-1) | 24 hours after first (pre-hospital) dose of study drug
Laboratory analysis of t-PA/PAI-1 complexes | At the end of 8 hour infusion of study drug
  Substudy
Laboratory analysis of t-PA/PAI-1 complexes | 24 hours after first (pre-hospital) dose of study drug
  Substudy
Laboratory analysis of thrombin activatable fibrinolysis inhibitor (TAFI) | At the end of 8 hour infusion of study drug
  Substudy
Laboratory analysis of thrombin activatable fibrinolysis inhibitor (TAFI) | 24 hours after first (pre-hospital) dose of study drug
  Substudy
Laboratory analysis of interleukins (IL-2, IL-4, IL-6, IL-8, IL-10) | At the end of 8 hour infusion of study drug
  Substudy
Laboratory analysis of interleukins (IL-2, IL-4, IL-6, IL-8, IL-10) | 24 hours after first (pre-hospital) dose of study drug
  Substudy
Laboratory analysis of granulocyte macrophage colony-stimulating factor (GM-CSF) | At the end of 8 hour infusion of study drug
  Substudy
Laboratory analysis of granulocyte macrophage colony-stimulating factor (GM-CSF) | 24 hours after first (pre-hospital) dose of study drug
  Substudy
Laboratory analysis of interferon gamma | At the end of 8 hour infusion of study drug
  Substudy
Laboratory analysis of interferon gamma | 24 hours after first (pre-hospital) dose of study drug
  Substudy
Laboratory analysis of tumour necrosis factor alpha | At the end of 8 hour infusion of study drug
  Substudy
Laboratory analysis of tumour necrosis factor alpha | 24 hours after first (pre-hospital) dose of study drug
  Substudy
TXA concentration in blood | 8 hours after first dose of study drug
  substudy
TXA concentration in blood | 24 hours after first dose of study drug
  substudy

CONTACTS AND LOCATIONS:
Overall Officials: Russell L Gruen, MBBS PhD, Principal Investigator — Monash University
Locations (33):
- Australia (26):
  - Lismore Base Hospital, Lismore, New South Wales
  - NNSW Medical Retrieval Service, Lismore, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - CareFlight, Northmead, New South Wales
  - Orange Base Hospital, Orange, New South Wales
  - Ambulance Service of New South Wales, Rozelle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Wagga Wagga Base Hospital, Wagga Wagga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - St John Ambulance, Darwin, Northern Territory
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Gold Coast Hospital, Gold Coast, Queensland
  - Queensland Ambulance Service, Kedron, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - South Australia Ambulance Service, Eastwood, South Australia
  - Ambulance Tasmania, Hobart, Tasmania
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ambulance Victoria, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St John Ambulance Western Australia, Geraldton, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (7):
  - St John Ambulance, Albany
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Waikato Hospital, Hamilton West
  - Hawke's Bay, Hastings
  - Wellington Free Ambulance, Wellington
  - Wellington Hospital, Wellington

REFERENCES:
- [Background] Gruen RL, Jacobs IG, Reade MC; PATCH-Trauma study. Trauma and tranexamic acid. Med J Aust. 2013 Sep 2;199(5):310-1. doi: 10.5694/mja13.10747. No abstract available. PMID 23992173
- [Background] Reade MC, Pitt V, Gruen RL. Tranexamic acid and trauma: current status and knowledge gaps with recommended research priorities. Shock. 2013 Aug;40(2):160-1. doi: 10.1097/SHK.0b013e31829ab240. No abstract available. PMID 23860584
- [Background] Mitra B, Mazur S, Cameron PA, Bernard S, Burns B, Smith A, Rashford S, Fitzgerald M, Smith K, Gruen RL; PATCH-Trauma Study Investigators. Tranexamic acid for trauma: filling the 'GAP' in evidence. Emerg Med Australas. 2014 Apr;26(2):194-7. doi: 10.1111/1742-6723.12172. PMID 24708011
- [Background] Gruen RL, Mitra B. Tranexamic acid for trauma. Lancet. 2011 Mar 26;377(9771):1052-4. doi: 10.1016/S0140-6736(11)60396-6. No abstract available. PMID 21439636
- [Background] Mitra B, Cameron PA, Mori A, Maini A, Fitzgerald M, Paul E, Street A. Early prediction of acute traumatic coagulopathy. Resuscitation. 2011 Sep;82(9):1208-13. doi: 10.1016/j.resuscitation.2011.04.007. Epub 2011 Apr 21. PMID 21600687
- [Derived] Mitra B, Reade MC, Bernard S, Dicker B, Maegele M, Gruen RL. High ratio of plasma to red cells in contemporary resuscitation of haemorrhagic shock after trauma: a secondary analysis of the PATCH-trauma trial. Scand J Trauma Resusc Emerg Med. 2025 Oct 2;33(1):154. doi: 10.1186/s13049-025-01476-2. PMID 41039456
- [Derived] PATCH-Trauma Investigators and the ANZICS Clinical Trials Group; Gruen RL, Mitra B, Bernard SA, McArthur CJ, Burns B, Gantner DC, Maegele M, Cameron PA, Dicker B, Forbes AB, Hurford S, Martin CA, Mazur SM, Medcalf RL, Murray LJ, Myles PS, Ng SJ, Pitt V, Rashford S, Reade MC, Swain AH, Trapani T, Young PJ. Prehospital Tranexamic Acid for Severe Trauma. N Engl J Med. 2023 Jul 13;389(2):127-136. doi: 10.1056/NEJMoa2215457. Epub 2023 Jun 14. PMID 37314244
- [Derived] Mitra B, Bernard S, Gantner D, Burns B, Reade MC, Murray L, Trapani T, Pitt V, McArthur C, Forbes A, Maegele M, Gruen RL; PATCH-Trauma study investigators; PATCH-Trauma Study investigators. Protocol for a multicentre prehospital randomised controlled trial investigating tranexamic acid in severe trauma: the PATCH-Trauma trial. BMJ Open. 2021 Mar 15;11(3):e046522. doi: 10.1136/bmjopen-2020-046522. PMID 33722875
- See also: PATCH study website — http://patchtrauma.org